CLINICAL TRIAL: NCT02452762
Title: Rapid Normalization of Vitamin D in Critically Ill Children: A Phase II Dose Evaluation Randomized Controlled Trial
Acronym: VITdAL-PICU
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Children's Hospital of Eastern Ontario (Other)
Responsible Party: Principal Investigator, James Dayre McNally, Pediatric Intensivist, Children's Hospital of Eastern Ontario
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VITdAL-PICU-01
Record Dates: First submitted 2015-05-15; First posted 2015-05-25 (Estimated); Results first posted 2021-08-13 (Actual); Last update posted 2021-08-13 (Actual); Status verified 2021-07

CONDITIONS: Hypovitaminosis D
MeSH Terms: conditions — Vitamin D Deficiency | interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Enteral Loading Arm (Experimental): Vitamin D3 (cholecalciferol) - Single dose at enrolment of 10000 IU/kg of cholecalciferol (max 400000 IU)
  Interventions: Drug: Vitamin D3
- Placebo Arm (Placebo Comparator): Patients will receive a placebo solution equivalent in volume to the dose of cholecalciferol administered to patients in the enteral loading arm.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Vitamin D3
  Other Names: Cholecalciferol
  Arms: Enteral Loading Arm
Drug: Placebo
  Arms: Placebo Arm

SUMMARY:
Documented roles for vitamin D in calcium homeostasis, cardiovascular and respiratory health, inflammation, innate immunity, and neuromuscular function have led to the hypothesis that deficiency might represent a modifiable risk factor for outcomes in critical illness. In recent years, dozens of adult studies have reported both high deficiency rates, and associations between lower vitamin D levels and organ dysfunction, health resource utilization, and mortality in the intensive care unit (ICU). More recently, similar observations have been made in critically ill pediatric populations. The cumulative body of basic science and clinical literature demonstrates that deficiency is common in critical illness and rapid normalization of vitamin D status could improve clinical outcomes and/or reduce health care costs. However, before conducting a phase III trial to determine whether restoration of vitamin D status improves outcomes in the PICU, the appropriate dosing regimen must be identified. Consequently, the investigators propose a phase II, double blind randomized controlled trial to determine a loading therapy dosing regimen that can safely and rapidly normalize vitamin D status in critically ill children.

DETAILED DESCRIPTION:
Background & Rationale: Documented roles for vitamin D in calcium homeostasis, cardiovascular and respiratory health, inflammation, innate immunity, and neuromuscular function have led to the hypothesis that deficiency might represent a modifiable risk factor for outcomes in critical illness. In recent years, dozens of adult studies have reported both high deficiency rates, and associations between lower vitamin D levels and organ dysfunction, health resource utilization, and mortality in the intensive care unit (ICU). More recently, similar observations have been made in critically ill pediatric populations. The cumulative body of basic science and clinical literature demonstrates that deficiency is common in critical illness and rapid normalization of vitamin D status could improve clinical outcomes and/or reduce health care costs. However, before conducting a phase III trial to determine whether restoration of vitamin D status improves outcomes in the PICU, the appropriate dosing regimen must be identified. Consequently, the investigators propose a phase II, double blind randomized controlled trial to determine a loading therapy dosing regimen that can safely and rapidly normalize vitamin D status in critically ill children.

Objectives:

Primary Objective: Determine whether a weight-based loading protocol can rapidly normalize blood vitamin D levels in critically ill children Secondary Objectives: (1) Evaluate whether a weight-based loading protocol, when compared with usual care, results in a greater occurrence of vitamin D related adverse events (hypercalcemia, hypercalciuria); and (2) determine the barriers to and feasibility of a multicenter phase III randomized control trial evaluating whether rapid vitamin D normalization improves clinical outcome and/or reduces health care spending in critically ill children.

Eligibility Criteria: The inclusion criteria for this study are: (i) Admitted to ICU, (ii) Corrected gestational age > 37 weeks to age < 18 years, (iii) Expected ICU admission in excess of 48 hours and expected access for blood work at Day 7 of hospital admission, and (iv) Blood 25(OH)D less than 50 nmol/L (regardless of prior approach to supplementation). Exclusion criteria are: (i) Significant gastrointestinal disorder preventing enteral drug administration (e.g. necrotizing enterocolitis); (ii) Hypercalcemia (excluding transient abnormalities and those related to parenteral calcium administration for hypocalcemia); (iii) Confirmed or suspected William's syndrome; (iv) Patient known to have nephrolithiasis or Nephrocalcinosis; (v) Imminent plan for withdrawal of care or transfer to another ICU; (vi) Physician refusal; (vii) Previous enrollment in the study; (viii) Patient known to have granulomatous disease (tuberculosis or sarcoidosis), (ix) Severe liver dysfunction/liver failure; (x) Patient know to have hypersensitivity or allergy to vitamin D or any of the non-medicinal ingredients of the formulation; (xi) Patient on thiazide diuretics who is also receiving regular ongoing calcium supplementation above the daily recommended intake (for reasons other than hypocalcemia); (xii) Adolescent female of child-bearing age with a positive serum pregnancy test; or (xiii) Patient on digoxin-therapy

Patients meeting inclusion criteria #1-3 and with no exclusion criteria will be approached regarding participation. If consent is given, 25OHD will be determined and those under 50 nmol/L will be randomized. Participants will be stratified by age in two categories (above 30 days of age or below/equal to 30 days of age). Randomization/allocation concealment will be performed using a web-based randomization system.

Interventions: All participants may also receive standard vitamin D dosing (e.g. 400 IU/day). Sixty-seven patients will be randomized 2:1 to the intervention (Enteral loading arm)

1. Enteral loading arm: 10000 IU/kg of cholecalciferol (max 400000 IU)
2. Placebo arm: For blinding purposes, this arm will receive a placebo solution

Data Collection: Blood and urine will be collected on days 0 (enrolment day), 1, 2, 3, 7, hospital discharge, and after interventions or triggers known to influence vitamin D status (e.g. cardiopulmonary bypass, hospital stay >30 days). Information on demographics, hospital course, adverse events, and health resource utilization will be entered into an electronic case report form.

Sample Size: Randomization of 40 children into the loading arm will provide sufficient power to estimate the proportion achieving target 25OHD with a confidence interval of ±15%. Assuming a 5% non-compliance/drop-out rate in each arm, randomization of 60 patients (total) may be required to achieve the desired power. The dosing regimen for this study was changed from a double dose to a single dose after the first seven patients were enrolled. As a result, the sample size was increased to 67 patients. All patients (n=67) will be included in the final intention to treat analysis. The 60 patients who received a single dose will be included in the per protocol analysis.

Significance: Critical illness occurs in tens of thousands of children each year in North America and can result in death, significant suffering, prolonged periods of rehabilitation, and chronic illness. High vitamin D deficiency rates in PICUs and the recognized interaction between vitamin D status and the health of multiple organ systems suggest that vitamin D could represent an inexpensive, safe means of improving outcomes and reducing health care spending. Unfortunately, approved daily dosing regimens require months to restore vitamin D levels and there have been no studies of loading therapy in pediatric critical illness. Consequently, despite significant literature suggesting vitamin D deficiency to be a modifiable risk factor, there is no evidence to inform physicians on the true benefits or risks of loading therapy. The proposed phase II clinical trial will determine how to provide cholecalciferol loads to facilitate rapid normalization of vitamin D levels, and provide initial information on toxicity.

ELIGIBILITY:
Inclusion Criteria:

(i) Admitted to ICU; (ii) Corrected gestational age > 37 weeks to age < 18 years; (iii) Expected ICU admission in excess of 48 hours and expected access for blood work at Day 7 of hospital admission; (iv) Blood 25OHD less than 50 nmol/L (regardless of prior approach to supplementation)

Exclusion Criteria:

(i) Significant gastrointestinal disorder preventing enteral drug administration (e.g. necrotizing enterocolitis); (ii) Hypercalcemia (excluding transient abnormalities and those related to parenteral calcium administration for hypocalcemia); (iii) Confirmed or suspected William's syndrome; (iv) Patient known to have nephrolithiasis or Nephrocalcinosis; (v) Imminent plan for withdrawal of care or transfer to another ICU; (vi) Physician refusal; (vii) Previous enrollment in the study; (viii) Patient known to have granulomatous disease (tuberculosis or sarcoidosis), (ix) Severe liver dysfunction/liver failure; (x) Patient know to have hypersensitivity or allergy to vitamin D or any of the non-medicinal ingredients of the formulation; (xi) Patient on thiazide diuretics who is also receiving regular ongoing calcium supplementation above the daily recommended intake (for reasons other than hypocalcemia); (xii) Adolescent female of child-bearing age with a positive serum pregnancy test; or (xiii) Patient on digoxin-therapy

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 67 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2017-11 (Actual); Study Completion 2018-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James D McNally, Principal Investigator — Children's Hospital of Eastern Ontario; Menon Kusum, Study Chair — Children's Hospital of Eastern Ontario; McIntyre Lauralyn, Study Chair — The Ottawa Hospital; Fergusson Dean, Study Chair — The Ottawa Hospital; Amrein Karin, Study Chair — Medical University of Graz
Locations (4):
- Medical University of Graz, Graz, Austria
- Canada (2):
  - Division of Critical Care, Department of Pediatrics, Victoria Hospital, London, Ontario
  - Children's Hospital of Eastern Ontario, Ottawa, Ontario
- Hospital Guillermo Grant Benavente, Concepción, Chile

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] O'Hearn K, Menon K, Weiler HA, Amrein K, Fergusson D, Gunz A, Bustos R, Campos R, Catalan V, Roedl S, Tsampalieros A, Barrowman N, Geier P, Henderson M, Khamessan A, Lawson ML, McIntyre L, Redpath S, Jones G, Kaufmann M, McNally D; Canadian Critical Care Trials Group. A phase II dose evaluation pilot feasibility randomized controlled trial of cholecalciferol in critically ill children with vitamin D deficiency (VITdAL-PICU study). BMC Pediatr. 2023 Aug 14;23(1):397. doi: 10.1186/s12887-023-04205-9. PMID 37580663
- [Derived] McNally D, Amrein K, O'Hearn K, Fergusson D, Geier P, Henderson M, Khamessan A, Lawson ML, McIntyre L, Redpath S, Weiler HA, Menon K; Canadian Critical Care Trials Group. Study protocol for a phase II dose evaluation randomized controlled trial of cholecalciferol in critically ill children with vitamin D deficiency (VITdAL-PICU study). Pilot Feasibility Stud. 2017 Dec 8;3:70. doi: 10.1186/s40814-017-0214-z. eCollection 2017. PMID 29234503

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Eligible participants were recruited from participating PICUs and one Neonatal Intensive Care Unit (NICU) between January 2016 to August 2017
Pre-assignment Details: This study did not involve a wash out or run-in period. The trial intervention initially involved two doses of study drug (placebo or cholecalciferol): i) At time of enrollment, and i) a day 3 dose dependent on the 25(OH)D concentration achieved. However, after randomization of the first 12 patients the intervention was adjusted to a single-dose protocol. Seven children who were enrolled under the two-dose protocol received >1 loading dose of cholecalciferol and were excluded from the analysis.
Groups:
- Enteral Loading Arm: Vitamin D3 (cholecalciferol) - Single dose at enrolment of 10000 IU/kg of cholecalciferol (max 400000 IU)
  Vitamin D3
- Placebo Arm: Patients will receive a placebo solution equivalent in volume to the dose of cholecalciferol administered to patients in the enteral loading arm.
  Placebo
Period: Overall Study
Arm/Group | Enteral Loading Arm | Placebo Arm
Started | 45 | 22
Completed | 40 | 19
Not Completed | 5 | 3
Not completed — Received >1 loading dose of cholecalciferol and analyzed separately | 4 | 3
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Enteral Loading Arm | Placebo Arm | Total
Number analyzed (Participants) | 40 | 19 | 59
Age, Continuous [Median (Inter-Quartile Range); unit: Months] | 13.4 [2.1 to 86.6] | 11.8 [2.1 to 87.9] | 12.8 [2.0 to 87.1]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 9 | 25
  Male | 24 | 10 | 34
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Canada | 33 | 16 | 49
  Austria | 1 | 1 | 2
  Chile | 6 | 2 | 8
Mechanical ventilation required, frequency [Count of Participants; unit: Participants] | 32 | 16 | 48
Received catecholamines, frequency [Count of Participants; unit: Participants] | 20 | 9 | 29
ICU type, frequency [Count of Participants; unit: Participants]
  Pediatric Intensive Care Unit | 37 | 17 | 54
  Neonatal Intensive Care Unit | 3 | 2 | 5
ICU Admission season, frequency [Count of Participants; unit: Participants]
  Fall | 8 | 4 | 12
  Winter | 11 | 7 | 18
  Spring | 9 | 4 | 13
  Summer | 12 | 4 | 16

OUTCOME MEASURES:

1. Primary Outcome: Vitamin D Status
Description: The percentage of critically ill children who achieve a blood 25OHD concentration above 75 nmol/L by day 7
Time Frame: 7 days
Population: A blood sample for the primary outcome analysis was available for 56 participants, 38 in the treatment arm and 18 in the placebo arm.
Measure: Number (95% Confidence Interval); unit: Percentage of participants in study arm
Arm/Group | Enteral Loading Arm | Placebo Arm
Number analyzed (Participants) | 38 | 18
Percentage of participants in study arm | 81.6 [66.6 to 90.8] | 5.6 [1.0 to 25.8]

2. Secondary Outcome: Patient Accrual Rate
Description: The investigators will determine the feasibility of a subsequent multicentre phase III interventional study through an evaluation of patient accrual rate. The expected patient accrual rate is 88 patients over a 2-year period (2-5 patients per month per centre; low estimate 60 patients (0-2 per month per centre). The study will be considered feasible if the patient accrual rate is achieved
Time Frame: 2 years
Population: The number of patients per enrolled per month per centre
Measure: Number; unit: Number of patients enrolled per month
Groups:
- Overall Cohort: Includes all randomized participants (both the Enteral Loading Arm and the Placebo Arm)
Arm/Group | Overall Cohort
Number analyzed (Participants) | 67
Number of patients enrolled per month | 3.35

3. Secondary Outcome: Vitamin D Related Adverse Events
Description: A measurable difference in clinically significant adverse events between the loading dose and placebo arms in unlikely in a phase II study. Therefore, the investigators will evaluate for potential toxicity using two well accepted surrogate outcome measures: (1) Hypercalcemia - The investigators will define hypercalcemia as an ionized calcium level above 1.40 mmol/L (children under 8 weeks as > 1.45 mmol/l); and (2) Hypercalciuria - Hypercalciuria will be defined as an elevated calcium:creatinine ratio above age-based normal values
Time Frame: On days 1, 2, 3, 7, hospital discharge (expected average of 2 weeks)
Measure: Count of Participants; unit: Participants
Arm/Group | Enteral Loading Arm | Placebo Arm
Number analyzed (Participants) | 40 | 19
Participants
  Hypercalcemia | 0 | 0
  Hypdercalciuria | 6 | 4
  No Hypercalcemia or Hypercaliuria | 34 | 15

4. Secondary Outcome: Vitamin D Axis Function - Calcium
Description: Improved signalling through the vitamin D axis will be evaluated through an evaluation of blood calcium levels (i.e. calcium metabolism). Calcium levels will be reported as median plus interquartile range and will be compared between the 2 study groups.
Time Frame: On day 0, 3, 7, hospital discharge (expected average of 2 weeks)
Measure: Median (Inter-Quartile Range); unit: mmol/mmol
Arm/Group | Enteral Loading Arm | Placebo Arm
Number analyzed (Participants) | 40 | 19
mmol/mmol
  Day 0 - Lowest | 1.17 [1.13 to 1.2] | 1.18 [1.14 to 1.23]
  Day 0 - Highest | 1.22 [1.17 to 1.28] | 1.21 [1.17 to 1.29]
  Day 3 - Lowest ionized calcium concentration | 1.16 [1.06 to 1.26] | 1.12 [1.09 to 1.18]
  Day 3 - Highest ionized calcium concentration | 1.21 [1.15 to 1.29] | 1.27 [1.14 to 1.27]
  Day 7 - Lowest ionized calcium concentration | 1.17 [1.12 to 1.23] | 1.17 [1.10 to 1.19]
  Day 7 - Highest ionized calcium concentration | 1.22 [1.18 to 1.27] | 1.18 [1.17 to 1.30]
  Hospital discharge - Lowest ionized calcium concentration | 1.24 [1.18 to 1.32] | 1.20 [1.15 to 1.27]
  Hospital discharge - Highest ionized calcium concentration | 1.26 [1.18 to 1.32] | 1.24 [1.18 to 1.29]

5. Secondary Outcome: Vitamin D Axis Function - 1,25-dihydroxyvitamin D
Description: Improved signalling through the vitamin D axis will be evaluated through an evaluation of blood 1,25OHD levels. 1,25 levels will be reported as median plus interquartile range and will be compared between the 2 study groups.
Time Frame: On day 3, 7, hospital discharge (expected average of 2 weeks)
Population: Data was not collected for this outcome. Due to insufficient funding and insufficient blood sample volume after analysis of the primary outcome, we were unable to complete this analysis.
Arm/Group | Enteral Loading Arm | Placebo Arm
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Immune Function - Cathelicidin
Description: Immune function will be evaluated through an evaluation of blood cathelicidin levels. Cathelicidin levels will be reported as median plus interquartile range and will be compared between the 2 study groups.
Time Frame: On day 3, 7, hospital discharge (expected average of 2 weeks)
Population: as for outcome 5
Arm/Group | Enteral Loading Arm | Placebo Arm
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Participants were monitored for adverse events from the time of study enrollment (administration of the study drug) until 90 days following enrollment.
Description: Ionized calcium levels and urine calcium:creatinine ratios from study samples were monitored in real time by the site investigator for hypercalcemia (study days 1, 2, 3, 7 and at hospital discharge) and hypercalciuria (study day 3, 7 and at hospital discharge). Additionally, the 25(OH)D level at Day 7/discharge was reviewed by the study nephrologist
Arm/Group | Enteral Loading Arm | Placebo Arm
All-Cause Mortality (participants affected / at risk) | 3/40 | 2/19
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/19
Other Adverse Events (participants affected / at risk) | 6/40 | 4/19
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Enteral Loading Arm (N=40) | Placebo Arm (N=19)
Nephrocalcinosis (Investigations) | 0 (0) | 0 (0) — Nephrocalcinosis on abdominal ultrasound
Persistent hypercalcemia (Endocrine disorders) | 0 (0) | 0 (0) — Ionized blood calcium >1.4 mmol/mmol in children 2 months and older, or an ionized blood calcium >1.45 mmol/mmol in children younger than 2 months
Persistent hypercalciuria (Endocrine disorders) | 6 (6) | 4 (4) — Calcium:creatinine ratio above age-established thresholds in two, sequential post-intervention urine samples

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-08-23): https://cdn.clinicaltrials.gov/large-docs/62/NCT02452762/Prot_SAP_000.pdf